CLINICAL TRIAL: NCT04370158
Title: Interstitial Lung Diseases Cohort Study in China
Acronym: ILD-China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Collaborators: The First Affiliated Hospital of Guangzhou Medical University (Other); Xiangya Hospital of Central South University (Other); First Hospital of China Medical University (Other); The Fourth Affiliated Hospital of China Medical University (Other); Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Dai Huaping, Deputy Director of Center for Respiratory Diseases, China-Japan Friendship Hospital
Other Study IDs: ChinaJapanFH003
Record Dates: First submitted 2020-04-29; First posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Interstitial Lung Diseases
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples With DNA — Blood, BALF, lung tissue, fibroblast
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: disease history — Clinical progression and prognosis of patients with interstitial lung diseases

SUMMARY:
In this project, the clinical diagnosis of interstitial lung diseases was carried out for the population with suspected interstitial lung diseases selected from the community cohort, and the confirmed patients were included into the existing clinical cohort of interstitial lung diseases, forming an interstitial lung diseases special disease cohort consisting of 3,000 patients and corresponding matched control groups. According to characteristics of interstitial lung disease and the needs of National Key R&D Program of China, this study will formulate unified clinical follow-up strategy to do long-term standardized clinical follow-up in patients with interstitial lung disease. The detailed information for clinical diagnosis and treatment as well as biological samples were collected to identify disease phenotype and build the database and biological sample library for interstitial lung disease cohort study. This study aims to provide evidence for molecular classification, screening and validation of biomarkers as well as precise diagnosis and prevention in patients with interstitial lung disease.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosed IPF during the last 3 months based upon ATS/ERS/JRS/ALAT guidelines 2011
* Agree to sign the informed consent

Exclusion Criteria:

* Lung transplantation expected within the next 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from the hospitals involved in this study
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Database and biological sample library for Chinese patients with interstitial lung disease | up to 4 years
  Data analyses will be mainly descriptive.

CONTACTS AND LOCATIONS:
Locations (1):
- Huaping Dai, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang H, Liu A, Ni Y, Wang J, Du J, Xi L, Qiang Y, Xie B, Ren Y, Wang S, Geng J, Deng Y, Huang S, Zhang R, Liu M, Dai H; China Interstitial Lung Disease Collaboration Network. Developing and Validation of a Multimodal-Based Machine Learning Model for Diagnosis of Usual Interstitial Pneumonia: A Prospective Multicenter Study. Chest. 2025 Sep 16:S0012-3692(25)05248-1. doi: 10.1016/j.chest.2025.08.034. Online ahead of print. PMID 40967367